CLINICAL TRIAL: NCT03256695
Title: A 12-Week, Open-Label Study to Evaluate the Relationship Between Use of Albuterol eMDPI, an Inhaled Short-Acting Beta Agonist "Rescue" Agent With an eModule, and Exacerbations in Patients (40 Years of Age or Older) With Chronic Obstructive Pulmonary Disease
Brief Title: Evaluate the Relationship Between Use of Albuterol Multidose Dry Powder Inhaler With an eModule (eMDPI) and Exacerbations in Participants With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABS-COPD-30065
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Results first posted 2019-08-06 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABS eMDPI (Experimental): Participants will receive 90 micrograms (mcg) of albuterol sulfate (ABS) via eMDPI (sitting on the upper part of the device for the purposes of detecting and storing usage information), 1 to 2 inhalations every 4 hours, as needed for 12 weeks. ABS eMDPI is a rescue/reliever agent that includes an eModule on top of the approved PROAIR RESPICLICK® inhaler. Participants will be allowed to continue use of other COPD and non-COPD medications as advised by their physician without changes unless deemed necessary by their physician.
  Interventions: Drug: Albuterol sulfate (ABS)

INTERVENTIONS:
Drug: Albuterol sulfate (ABS) — ABS will be administered via eMDPI as per the dose and schedule specified in the arm.

SUMMARY:
This is a Phase 3B, 12-week, multicenter, open-label study to evaluate the relationship between as-needed usage of albuterol eMDPI and Clinical Exacerbation-Chronic Obstructive Pulmonary Disease (CE-COPD) in adult participants at least 40 years of age with exacerbation-prone COPD.

ELIGIBILITY:
Inclusion Criteria:

* The participant has had at least 1 episode of moderate or severe CE-COPD over the past 12 months before screening.
* The participant must be able to demonstrate appropriate use of albuterol from the ABS eMDPI.
* The participant is currently using a short-acting beta agonist (SABA) reliever plus at least one of the following: long-acting beta agonist (LABA), an inhaled corticosteroid (ICS)/LABA, a long-acting muscarinic antagonist (LAMA), or a LABA/LAMA.
* The participant must be willing and able to comply with study requirements as specified in the protocol, including the use of a wearable accelerometer for the subset of participants who consent to use of the device.
* The participant is willing to discontinue all other rescue or maintenance SABA or antimuscarinic agents and replace them with the study-provided ABS eMDPI for the duration of the trial.
* Women of childbearing potential (not surgically sterile or greater than or equal to [≥]2 years postmenopausal) must have exclusively same-sex partners or use a highly effective method of birth control and must agree to continue the use of this method for the duration of the study and for 30 days after discontinuation of the investigational medicinal product (IMP).

  * Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* The participant has any clinically significant medical condition (treated or untreated) that, in the opinion of the investigator, would interfere with participation in the study.
* The participant has any other confounding underlying lung disorder other than COPD.
* The participant has used an investigational drug within 5 half-lives of it being discontinued or within1 month of Visit 2 (Baseline [Day 1]), whichever is longer.
* The participant is a pregnant or lactating woman, or plans to become pregnant during the study. Note: Any woman becoming pregnant during the study will be withdrawn from the study.
* The participant is known to be allergic to albuterol or any of the excipients in the IMP or rescue medication formulation (that is, lactose [milk protein]). Dietary lactose intolerance does not exclude the participant from inclusion in the study or as per the investigator's medical discretion.
* The participant has a history or presence of "silent" infections, including positive testing for human immunodeficiency virus types 1 and 2, hepatitis B, hepatitis C, and tuberculosis.

  * Additional criteria apply, please contact the investigator for more information.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (40):
- United States (40):
  - Teva Investigational Site 14682, Andalusia, Alabama
  - Teva Investigational Site 14704, Anniston, Alabama
  - Teva Investigational Site 14712, Mobile, Alabama
  - Teva Investigational Site 14702, Peoria, Arizona
  - Teva Investigational Site 14706, Gold River, California
  - Teva Investigational Site 14720, Waterbury, Connecticut
  - Teva Investigational Site 14725, Brandon, Florida
  - Teva Investigational Site 14711, Daytona Beach, Florida
  - Teva Investigational Site 14699, DeLand, Florida
  - Teva Investigational Site 14694, Edgewater, Florida
  - Teva Investigational Site 14701, Miami, Florida
  - Teva Investigational Site 14689, Miami, Florida
  - Teva Investigational Site 14678, Miami, Florida
  - Teva Investigational Site 14688, Orlando, Florida
  - Teva Investigational Site 14679, Valparaiso, Indiana
  - Teva Investigational Site 14677, North Dartmouth, Massachusetts
  - Teva Investigational Site 14705, Chesterfield, Missouri
  - Teva Investigational Site 14717, Omaha, Nebraska
  - Teva Investigational Site 14684, Toms River, New Jersey
  - Teva Investigational Site 14710, Charlotte, North Carolina
  - Teva Investigational Site 14696, Gastonia, North Carolina
  - Teva Investigational Site 14722, Greensboro, North Carolina
  - Teva Investigational Site 14692, Winston-Salem, North Carolina
  - Teva Investigational Site 14708, Columbus, Ohio
  - Teva Investigational Site 14703, Dayton, Ohio
  - Teva Investigational Site 14680, Grove City, Ohio
  - Teva Investigational Site 14709, Toledo, Ohio
  - Teva Investigational Site 14724, Willoughby, Ohio
  - Teva Investigational Site 14683, Pittsburgh, Pennsylvania
  - Teva Investigational Site 14681, Charleston, South Carolina
  - Teva Investigational Site 14686, Easley, South Carolina
  - Teva Investigational Site 14719, Gaffney, South Carolina
  - Teva Investigational Site 14691, Greenville, South Carolina
  - Teva Investigational Site 14695, Mt. Pleasant, South Carolina
  - Teva Investigational Site 14715, Spartanburg, South Carolina
  - Teva Investigational Site 14718, Spartanburg, South Carolina
  - Teva Investigational Site 14707, Union, South Carolina
  - Teva Investigational Site 14716, San Antonio, Texas
  - Teva Investigational Site 14713, Richmond, Virginia
  - Teva Investigational Site 14687, Spokane, Washington

REFERENCES:
- [Derived] Snyder LD, DePietro M, Reich M, Neely ML, Lugogo N, Pleasants R, Li T, Granovsky L, Brown R, Safioti G. Predictive machine learning algorithm for COPD exacerbations using a digital inhaler with integrated sensors. BMJ Open Respir Res. 2025 May 12;12(1):e002577. doi: 10.1136/bmjresp-2024-002577. PMID 40355297

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 423 participants with exacerbation-prone chronic obstructive pulmonary disease (COPD) were screened, of which 405 participants at 40 investigational centers in the United States met entry criteria and were considered to be eligible for enrollment into the study.
Groups:
- ABS eMDPI: Participants received 90 micrograms (mcg) of albuterol sulfate (ABS) via a multidose dry powder inhaler (MDPI) with an eModule (eMDPI) (that had a sensor on the top of device for the purposes of detecting and storing usage information), 1 to 2 inhalations every 4 hours, as needed for 12 weeks. ABS eMDPI was a rescue/reliever agent that included an eModule on top of the approved PROAIR RESPICLICK® inhaler. Participants were allowed to continue use of other COPD and non-COPD medications as advised by their physician without changes unless deemed necessary by their physician.
Period: Overall Study
Arm/Group | ABS eMDPI
Started | 405
Used ABS eMDPI at Least Once | 390
Completed | 366
Not Completed | 39
Not completed — Adverse Event | 8
Not completed — Death | 2
Not completed — Withdrawal by Subject | 14
Not completed — Non-compliance with study drug | 1
Not completed — Lost to Follow-up | 3
Not completed — Lack of Efficacy | 3
Not completed — Protocol Violation | 5
Not completed — Other than specified | 3

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all enrolled participants regardless of whether a participant took any investigational medicinal product (IMP).
Groups:
- ABS eMDPI: Participants received 90 mcg of ABS via eMDPI (that had a sensor on the top of device for the purposes of detecting and storing usage information), 1 to 2 inhalations every 4 hours, as needed for 12 weeks. ABS eMDPI was a rescue/reliever agent that included an eModule on top of the approved PROAIR RESPICLICK® inhaler. Participants were allowed to continue use of other COPD and non-COPD medications as advised by their physician without changes unless deemed necessary by their physician.
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 405
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220
  Male | 185
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34
  Not Hispanic or Latino | 371
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 38
  White | 365
  More than one race | 0
  Unknown or Not Reported | 0
Number of COPD Exacerbations in the Past 12 Months [Mean (Standard Deviation); unit: exacerbations] | 1.5 (0.98)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Exacerbation of COPD (CE-COPD) Rate: Percentage of Participants Who Experienced at Least 1 Moderate or Severe CE-COPD
Description: CE-COPD was an occurrence of either severe CE-COPD or moderate CE-COPD. Severe CE-COPD was defined as an event that involved worsening respiratory symptoms for at least 2 consecutive days requiring treatment with systemic corticosteroids (SCS; at least 10 milligrams [mg] prednisone equivalent above baseline) and/or systemic antibiotics and a hospitalization for CE COPD.
  Moderate CE-COPD was defined as an event that involved worsening respiratory symptoms for at least 2 consecutive days requiring treatment with SCS (at least 10 mg prednisone equivalent above baseline), and/or systemic antibiotics, and an unscheduled encounter (such as a phone call, an office visit, an urgent care visit, or an emergency care visit) for a CE-COPD, but not a hospitalization.
Time Frame: Baseline (Day 1) to Week 12
Population: ITT analysis set included all enrolled participants regardless of whether a participant took any IMP. Participants with CE-COPD during study Day 1 through study Day 7 were excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 396
percentage of participants | 28

2. Primary Outcome: Total Number of Albuterol Inhalations in the Days Preceding the Symptom Peak of a CE-COPD Event
Description: Severe CE-COPD: an event that involved worsening respiratory symptoms for at least 2 consecutive days requiring treatment with SCS (at least 10 mg prednisone equivalent above baseline) and/or systemic antibiotics and a hospitalization. Moderate CE-COPD: an event that involved worsening respiratory symptoms for at least 2 consecutive days requiring treatment with SCS (at least 10 mg prednisone equivalent above baseline), and/or systemic antibiotics, and an unscheduled encounter (such as a phone call, office visit, urgent care visit, or emergency care visit), but not a hospitalization. Total number of inhalations taken in 1 day(24-hour period on day prior to date of CE-COPD symptom peak) and at 3,5,7,10,14, and 21 days preceding the date of CE-COPD symptom peak were reported. If a participant experienced multiple CE-COPD events, number of inhalations preceding symptom peak of a subsequent event was counted since end of previous event. Average of inhalations of all events were presented.
Time Frame: Baseline to Week 12
Population: ITT analysis set:all enrolled participants regardless of whether a participant took any IMP. Participants with CE-COPD during Day 1 to Day 7 were excluded. 'Overall number of participants analyzed'= participants experiencing at least 1 moderate or severe CE-COPD.
Measure: Mean (Standard Deviation); unit: inhalations
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 109
inhalations
  Day 1 prior to CE-COPD symptom peak | 3.7 (4.36)
  Day 3 prior to CE-COPD symptom peak | 3.5 (4.61)
  Day 5 prior to CE-COPD symptom peak | 4.2 (5.35)
  Day 7 prior to CE-COPD symptom peak | 3.4 (4.45)
  Day 10 prior to CE-COPD symptom peak | 3.2 (4.41)
  Day 14 prior to CE-COPD symptom peak | 3.4 (4.42)
  Day 21 prior to CE-COPD symptom peak | 3.1 (4.54)

3. Primary Outcome: Number of Days Prior to the Symptom Peak of a CE-COPD Event When Albuterol Use Increased
Description: CE-COPD: occurrence of moderate or severe CE-COPD. Severe CE-COPD: an event that involved worsening respiratory symptoms for at least 2 consecutive days requiring treatment with SCS (at least 10 mg prednisone equivalent above baseline) and/or systemic antibiotics and a hospitalization. Moderate CE-COPD: an event that involved worsening respiratory symptoms for at least 2 consecutive days requiring treatment with SCS (at least 10 mg prednisone equivalent above baseline), and/or systemic antibiotics, and an unscheduled encounter (such as a phone call, an office visit, an urgent care visit, or an emergency care visit), but not a hospitalization. Number of days of increased albuterol use prior to the symptom peak of a CE-COPD was reported for first increase of daily albuterol use; 2 and 4 inhalations in a single day from baseline. increased daily albuterol use was defined as single-day increase of greater than (>) 20 percent (%) from baseline.
Time Frame: Baseline to Week 12
Population: ITT analysis set: all enrolled participants regardless of whether a participant took any IMP. 'Overall number of participants analyzed'= participants experiencing at least 1 moderate or severe CE-COPD. 'Number analyzed'=participants evaluable for specified categories. Participants with CE-COPD during Day 1 to Day 7 were excluded.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 109
days
  Days from albuterol use >20% increase to CE-COPD: number analyzed (Participants) | 96
  Days from albuterol use >20% increase to CE-COPD | 32.7 (19.92)
  Days from 2 inhalations increase to CE-COPD: number analyzed (Participants) | 66
  Days from 2 inhalations increase to CE-COPD | 31.2 (21.30)
  Days from 4 inhalations increase to CE-COPD: number analyzed (Participants) | 50
  Days from 4 inhalations increase to CE-COPD | 30.4 (21.24)

4. Primary Outcome: Number of Albuterol Uses in the 24 Hours Preceding a CE-COPD
Description: CE-COPD referred to occurrence of moderate or severe CE-COPD. Severe CE-COPD was defined as an event that involved worsening respiratory symptoms for at least 2 consecutive days requiring treatment with SCS (at least 10 mg prednisone equivalent above baseline) and/or systemic antibiotics and a hospitalization for CE COPD. Moderate CE-COPD was defined as an event that involved worsening respiratory symptoms for at least 2 consecutive days requiring treatment with SCS (at least 10 mg prednisone equivalent above baseline), and/or systemic antibiotics, and an unscheduled encounter (such as a phone call, an office visit, an urgent care visit, or an emergency care visit) for a CE-COPD, but not a hospitalization. Number of albuterol inhalations used in the 24 hours preceding a moderate or severe CE-COPD was reported.
Time Frame: Baseline to Week 12
Population: ITT analysis set: all enrolled participants regardless of whether a participant took any IMP. Participants with CE-COPD during Day 1 to Day 7 were excluded. 'Overall number of participants analyzed' = participants who experienced at least 1 moderate or severe CE-COPD and reported albuterol use in the 24 hours preceding a moderate or severe CE-COPD.
Measure: Mean (Standard Deviation); unit: inhalations/24 hours
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 109
inhalations/24 hours | 3.7 (4.36)

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by investigator. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: Baseline up to Week 12
Population: ITT analysis set included all enrolled participants regardless of whether a participant took any IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | ABS eMDPI
Number analyzed (Participants) | 405
Participants
  Any AEs | 190
  Severe AEs | 43
  Treatment-related AEs | 2
  Treatment-related severe AE | 0
  Serious AEs | 44
  AEs leading to discontinuation from study | 8
  CE-COPD related AEs | 118
  Device-related AEs | 0
  AEs leading to death | 2

ADVERSE EVENTS:
Time Frame: AEs were collected from signature of the informed consent form (ICF) to Week 12.
Description: AEs were reported from Baseline (Day 1) up to Week 12. ITT analysis set included all enrolled participants regardless of whether a participant took any IMP.
Arm/Group | ABS eMDPI
All-Cause Mortality (participants affected / at risk) | 2/405
Serious Adverse Events (participants affected / at risk) | 44/405
Other Adverse Events (participants affected / at risk) | 94/405
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABS eMDPI (N=405)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Osteomyelitis acute (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Pneumonia staphylococcal (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Burns first degree (Injury, poisoning and procedural complications) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1)
Influenza B virus test positive (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Substance use disorder (Psychiatric disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 22 (24)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABS eMDPI (N=405)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 94 (104)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT03256695/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT03256695/SAP_001.pdf